CLINICAL TRIAL: NCT04609865
Title: Impact of Intravenous Lidocaine on Clinical Outcomes of Patients With ARDS During COVID-19 Pandemia
Acronym: LidoCovid
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: departure of the principal investigator and inclusion difficulties
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7820
Record Dates: First submitted 2020-10-23; First posted 2020-10-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS); COVID-19; Corona Virus Infection
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19; Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine 2% (Experimental): The lidocaine infusion protocol is a bolus of 1 mg/kg (ideal weight), followed by 3mg/kg/h for the first hour, 1.5 mg/kg/h for the second hour, 0.72 mg/kg/h for the next 22 hours,and then 0.6mg/kg/h for 14 days or until extubation.
  Interventions: Drug: Lidocaine 2%
- Control (Placebo Comparator): The NaCl 0,9% infusion protocol is a bolus of 0.05 ml/kg (ideal weight), followed by 0.15 ml/kg/h for the first hour, 0.075 ml/kg/h for the second hour, 0.36 ml/kg/h for the next 22 hours, and then 0.03 ml/kg/h for 14 days or until extubation.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Lidocaine 2% — the lidocaine infusion protocol is a bolus of 1 mg/kg (ideal weight), followed by 3mg/kg/h for the first hour, 1.5 mg/kg/h for the second hour, 0.72 mg/kg/h for the next 22 hours, and then 0.6mg/kg/h for 14 days or until extubation.
  Arms: Lidocaine 2%
Drug: Control — The NaCl 0,9% infusion protocol is a bolus of 0.05 ml/kg (ideal weight), followed by 0.15 ml/kg/h for the first hour, 0.075 ml/kg/h for the second hour, 0.36 ml/kg/h for the next 22 hours, and then 0.03 ml/kg/h for 14 days or until extubation.
  Arms: Control

SUMMARY:
The purpose of our prospective monocentric, randomized, controlled trial is to evaluate the effects of intravenous lidocaine on gas exchange and inflammation in acute respiratory distress syndrome (ARDS) due or not to Covid-19 pneumonia.

Half of the patients will receive intravenous lidocaine and the other half will receive intravenous NaCl 0,9 % as placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Hospitalized in ICU
* Presence of all of the following conditions, within one week of a clinical insult or new or worsening respiratory symptoms:
* PaO2/FiO2 <300 mmHg with positive end-expiratory pressure (PEEP) ≥5 cmH2O
* Bilateral opacities not fully explained by cardiac failure or fluid overload
* Intubated and sedated for mechanical protective ventilation
* Affiliation to the French Sociale security
* Beta HCG negative for women

For Covid-19 subgroup:

- Covid-19 infection (RT-PCR < 7 days and/or another approved diagnostic technique and/or typical CT appearance of COVID-19 pneumonia

Exclusion Criteria:

* Allergy to amide local anesthetics
* Acute porphyria
* Disorders of atrioventricular conduction requiring a non-done permanent electrosystolic pacing
* Uncontrolled epilepsy
* Fluvoxamine treatment
* Class III antiarrythmic agent treatments (amiodarone, dronedarone)
* Class I antiarythmic agent (quinidine, disopyramide, hydroquinidine, flecainid, propafenone)
* Hepatocellular insufficiency defined by PT<15% in the absence of anti-vitamin K
* Patient under a tutelage measure or placed under judicial protection
* Known pregnancy
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
alveolar-capillary gas exchange after two days of treatment | At 48 hours after the first treatment administration
  PaO2/FiO2 ratio

SECONDARY OUTCOMES:
alveolar-capillary gas exchange From day 0 to day 21 or until coming out of intensive care | From day 0 to day 21 or until coming out of intensive care
  PaO2/FiO2 ratio : a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
Ventilator-free days | At day 28 and at day 90
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
Measure the effects of Intravenous Lidocaine on Biomarkers : Ferritin | At Day 0, day 2, day 7, day 14 and at day 21
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
Measure the effects of Intravenous Lidocaine on Biomarkers : bicarbonates | At Day 0, day 2, day 7, day 14 and at day 21
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
Measure the effects of Intravenous Lidocaine on Biomarkers : CRP | At Day 0, day 2, day 7, day 14 and at day 21
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
Measure the effects of Intravenous Lidocaine on Biomarkers : LDH | At Day 0, day 2, day 7, day 14 and at day 21
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
Measure the effects of Intravenous Lidocaine on Biomarkers : IL-6 | At Day 0, day 2, day 7, day 14 and at day 21
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
Measure the effects of Intravenous Lidocaine on Biomarkers : Tropo HS | At Day 0, day 2, day 7, day 14 and at day 21
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
Measure the effects of Intravenous Lidocaine on Biomarkers : Triglycerides | At Day 0, day 2, day 7, day 14 and at day 21
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
Measure the effects of Intravenous Lidocaine on Biomarkers : CBC with lymphocytes count | At Day 0, day 2, day 7, day 14 and at day 21
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
Antithrombotic activity of Intravenous Lidocaine on platelets | At Day 0, day 2, day 7, day 14 and at day 21
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
Antithrombotic activity of Intravenous Lidocaine on ACT ratio | At Day 0, day 2, day 7, day 14 and at day 21
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
Antithrombotic activity of Intravenous Lidocaine on fibrinogen | At Day 0, day 2, day 7, day 14 and at day 21
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
Antithrombotic activity of Intravenous Lidocaine on D-Dimers | At Day 0, day 2, day 7, day 14 and at day 21
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
Antithrombotic activity of Intravenous Lidocaine on TEG | At Day 0, day 2, day 7, day 14 and at day 21
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
Antithrombotic activity of Intravenous Lidocaine on thromboembolic events | At Day 0, day 2, day 7, day 14 and at day 21
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
Plasma concentration of albumin and Lidocaine | 4 hours after first administration, at day 2, day 7, day 14 and at day 21
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
Search for hemodynamic dysfynction: Blood pressure measurement in mmHg | daily from day one to day 14
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
  Blood pressure in mmHg will be measured
Search for hemodynamic dysfynction: Cardiac frequency in beats per minute will be assessed | daily from day one to day 14
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
  Cardiac frequency in beats per minute will be assessed
Search for hemodynamic dysfynction: Sinus rythm will be assessed | daily from day one to day 14
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
  Sinus rythm will be assessed
Search for hemodynamic dysfynction: Vasopressors and inotropes drugs use will be reported | daily from day one to day 14
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
  Vasopressors and inotropes drugs use will be reported
Search for hemodynamic dysfynction: EKG : PR, QRS, QTc intervals in ms will be measured | daily from day one to day 14
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
  EKG : PR, QRS, QTc intervals in ms will be measured
ICU ileus: laxation response | daily from Day 0 to Day 28
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
Opioids, sedative and curare sparing effect (drugs dosage) | daily from Day 0 to Day 28
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
Evaluate the impact of Lidocaine IV on ICU outcomes : re-intubation | From Day0 to Day28 and at Day90
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
Evaluate the impact of Lidocaine IV on ICU outcomes : ICU length of stay | From Day0 to Day28 and at Day90
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
Evaluate the impact of Lidocaine IV on ICU outcomes : ICU complications | From Day0 to Day28 and at Day90
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.
Cough at extubation time or in the 24 hours after extubation or weaning from respiratory support (in case of tracheostomy) | extubation day
  a comparison will be made between Lidocaine and control groups in patients with acute respiratory distress syndrome (ARDS) due to Covid-19 and in patients with ARDS without Covid-19.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Hautepierre, Strasbourg, Bas-Rhin, France

REFERENCES:
- [Derived] Muller M, Lefebvre F, Harlay ML, Glady L, Becker G, Muller C, Aberkane O, Tawk M, Julians M, Romoli A, Hecketsweiler S, Schneider F, Pottecher J, Chamaraux-Tran TN. Impact of intravenous lidocaine on clinical outcomes of patients with ARDS during COVID-19 pandemia (LidoCovid): A structured summary of a study protocol for a randomised controlled trial. Trials. 2021 Feb 11;22(1):131. doi: 10.1186/s13063-021-05095-x. PMID 33573681